CLINICAL TRIAL: NCT04545411
Title: Effect of Glucagon Receptor Antagonism on Ketogenesis in SGLT-2i Treated Subjects With T1D
Brief Title: Combination GRA and SGLT-2i Treatment in Type 1 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: REMD Biotherapeutics, Inc. (Industry); Juvenile Diabetes Research Foundation (Other); The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Principal Investigator, Jeremy Pettus, MD, Clinical Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: UC-MEDJP-03
Record Dates: First submitted 2020-08-28; First posted 2020-09-11 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — dapagliflozin; volagidemab

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, double-blind, cross-over, multi-dose study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A (Active Comparator): Daily, Oral,10mg dapagliflozin in combination with Weekly, Subcutaneous, 35mg in 1mL solution REMD-477
  Interventions: Drug: Dapagliflozin 10 MG [Farxiga]; Drug: REMD-477
- Treatment B (Placebo Comparator): Daily, Oral,10mg dapagliflozin in combination with Weekly, Subcutaneous, 1mL solution Placebo
  Interventions: Drug: Dapagliflozin 10 MG [Farxiga]; Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10 MG [Farxiga] — 4-Week, double-blind, once daily oral 10mg dapagliflozin
Drug: REMD-477 — 4-Week, double-blind, once weekly subcutaneous injection with 35mg REMD-477 in 1mL solution.
  Arms: Treatment A
Drug: Placebo — 4-Week, double-blind, once weekly subcutaneous injection with placebo in 1mL solution.
  Arms: Treatment B

SUMMARY:
A pilot study for individuals with Type 1 Diabetes who are willing to add an SGLT-2i (Sodium-Glucose Cotransporter-2 Inhibitor) in combination with placebo or a GRA (Glucagon Receptor Antagonist) to their current diabetes treatment regimen. There will be 15 study visits over approximately 14 weeks in this cross-over study design. Treatment "A" consists of an SGLT-2i + GRA for 4 weeks and treatment "B" consists of an SGLT-2i + placebo for 4 weeks. All participants will complete both treatment "A" and treatment "B" with a 6-week washout period in between the treatments. Testing includes 3 insulin withdraw challenges, 3 muscle biopsies, 3 fat biopsies, 3 vascular ultrasounds along with blood collection and vitals.

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind, cross-over, multi-dose study designed to elicit pilot data for a larger project. To accomplish the specific aims proposed, a single clinical trial will be conducted in which a maximum of 12 subjects with T1D, who are otherwise healthy, will be treated with an oral SGLT-2i (Sodium-Glucose Cotransporter-2 Inhibitor), 10mg dapagliflozin taken daily in combination with a GRA (Glucagon Receptor Antagonist), 70mg REMD-477 subcutaneous injection once a week or placebo (subcutaneous injection to match the volume of REMD-477) once a week. There will be two treatments: Treatment "A" consists of an SGLT-2i + GRA for 4 weeks and Treatment "B" consists of an SGLT-2i + placebo for 4 weeks. Participants will be randomly assigned to either start with Treatment A or Treatment B for the first 4 weeks of treatment. After completing the first treatment group, participants will be washed off all study drug for 6 weeks. After the washout period, participants will complete 4 weeks of dosing with the opposite treatment they received during the first 4 weeks.

There will be 15 study visits as outlined below:

1. Screening - Complete medical history, physical exam, review current medications, height/weight, vital signs, ECG and fasting laboratory (blood and urine) tests.
2. Baseline 1 - Complete vitals, weight, physical exam, fasting blood collection, download CGM data, collect insulin usage, complete measurements of blood vessels using EndoPat and ultrasound, complete diabetes questionnaires, and complete fat and muscle biopsies.
3. Baseline 2 - Complete vitals, weight, fasting blood collection, insulin withdraw procedure and start first dose of study medications.
4. Visit 4 - Complete vitals, weight, dose 2 of REMD-477/Placebo, review CGM data and insulin dosing.
5. Visit 5 - Complete vitals, weight, dose 3 of REMD-477/Placebo, review CGM data and insulin dosing.
6. Visit 6 - Complete vitals, weight, dose 4 of REMD-477/Placebo, review CGM data and insulin dosing.
7. Repeat Measures 1 - Complete vitals, weight, physical exam, fasting blood collection, download CGM data, collect insulin usage, complete measurements of blood vessels using EndoPat and ultrasound, complete diabetes questionnaires, and complete fat and muscle biopsies.
8. Repeat Measures 2 - Complete vitals, weight, fasting blood collection, insulin withdraw procedure and begin wash-out of study medications.
9. Crossover Visit - Update medical history, complete physical exam, review of current medications, weight, vital signs, fasting laboratory (blood and urine) tests, collect insulin usage, download CGM data and start opposite doses of medication.
10. Visit 10 - Complete vitals, weight, dose 2 of REMD-477/Placebo, review CGM data and insulin dosing.
11. Visit 11 - Complete vitals, weight, dose 3 of REMD-477/Placebo, review CGM data and insulin dosing.
12. Visit 12 - Complete vitals, weight, dose 4 of REMD-477/Placebo, review CGM data and insulin dosing.
13. Final Measures 1 - Complete vitals, weight, physical exam, fasting blood collection, download CGM data, collect insulin usage, complete measurements of blood vessels using EndoPat and ultrasound, complete diabetes questionnaires, and complete fat and muscle biopsies.
14. Final Measures 2 - Complete vitals, weight, fasting blood collection, insulin withdraw procedure and review CGM data/insulin dosing for return to pre-baseline diabetes treatment.
15. Safety Follow-up - Complete vitals, physical exam, weight, and review CGM data/insulin dosing to verify diabetes treatment is stable.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 18 and 65 years old, inclusive, at the time of screening;
2. Females of non-child bearing potential must be ≥ 1 year post-menopausal or documented as being surgically sterile. Females of child bearing potential must agree to use two methods of contraception during the entire study and for an additional 3 months after the end of dosing with the investigational product;
3. Male subjects must be willing to use clinically acceptable method of contraception during the entire study and for an additional 6 months after the end of the treatment period;
4. Diagnosed with Type 1 diabetes based on clinical history or as defined by the current American Diabetes Association (ADA) criteria for > 5 years;
5. Treatment with a stable insulin regimen (< 1u/kg per day) for at least 8 weeks before screening with continuous subcutaneous insulin infusion (CSII) via an insulin pump;
6. Currently using a Continuous Glucose Monitoring (CGM) system
7. HbA1c ≤ 9 % at screening;
8. A minimum weight of 50kg;
9. eGFR ≥ 60 mL/min/1.73m²
10. Able to provide written informed consent approved by an Institutional Review Board (IRB).

Exclusion Criteria:

1. History of T2DM, maturity onset diabetes of the young (MODY), pancreatic surgery or chronic pancreatitis
2. Pancreas, pancreatic islet cells or renal transplant recipient
3. T1DM treatment with any other antihyperglycemic drug (e.g. metformin, alpha- glucosidase inhibitors, SGLT-2 inhibitors, pramlintide, inhaled insulin, pre-mixed insulins, etc.) within 30 days of run-in (visit 2)
4. Occurrence of severe hypoglycemia involving coma and/or seizure that required hospitalization or hypoglycemia-related treatment by an emergency physician or paramedic within 3 months prior to Visit 1 or Visit 2
5. Occurrence of DKA within 3 months prior to Visit 1 or Visit 2
6. Occurrence of symptomatic hypotension within 3 months prior to Visit 1 (Screen) or Visit 2
7. Occurrence of multiple genital mycotic infections within 6 months prior to Visit 1 (Screen) or Visit 2
8. Acute coronary syndrome (non-STEMI, STEMI and unstable angina pectoris), stroke or transient ischemic attack (TIA) within 3 months prior to Visit 1 or Visit 2
9. Indication of liver disease, defined by serum levels of either alanine transaminase (ALT), aspartate transaminase (AST), or alkaline phosphatase above 3 x upper limit of normal (ULN) at Visit 1
10. Current signs and symptoms of anemia accompanied by a hemoglobin laboratory value at or below 10.0 g/dL at screening.
11. Active eating disorders such as bulimia or anorexia nervosa
12. Body Mass Index (BMI) < 18.5 kg/m2 and/or weight less than 50kg;
13. Whole blood donation of 1 pint (500 mL) within 8 weeks prior to Screening. Donations of plasma, packed RBCs, platelets or quantities less than 500 mL are allowed at investigator discretion;
14. Treatment with systemic corticosteroids within 30 days of run-in (visit 2), or planned initiation of such therapy at Visit 1 or Visit 2. Inhaled or topical use of corticosteroids (e.g. for asthma/chronic obstructive pulmonary disease) is acceptable.
15. Medical history of bladder cancer or treatment for any cancer in the last five years prior to Visit 1. Resected basal cell carcinoma considered cured is exempted.
16. Women who are pregnant, nursing, or who plan to become pregnant while in the trial
17. Intake of an investigational drug in another trial within 30 days prior to Visit 1
18. Patient not able to understand and comply with study requirements, based on Investigator's judgment
19. Any other clinical condition that, based on Investigator's judgment, would jeopardize patient safety during trial participation or would affect the study outcome (e.g. immunocompromised patients who might be at higher risk of developing genital or mycotic infections, patients with chronic viral infections etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Beta-hydroxybutyrate (BHB) Level | 4-Weeks
  The change from baseline in peak BHB production as measured by the insulin withdrawal challenge.
Change in Glycemic Control | 4-Weeks
  The change from baseline glycemic control as measured by a 2-week average of CGM "time-in-range".
Change in Glycemic Control | 4-Weeks
  The change from baseline glycemic control as measured by HbA1c.
Change in Vascular Endothelial Function | 4-Weeks
  The change from baseline in vascular endothelial function as measured by flow mediated dilation (brachial artery diameter).
Change in Vascular Endothelial Function | 4-Weeks
  The change from baseline in vascular endothelial function as measured by reactive hyperemia-peripheral arterial tonometry (reactive hyperemia index).

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego Altman Clinical & Translational Research Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No